CLINICAL TRIAL: NCT00197847
Title: Infection Surveillance in Intensive Care Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Herlev Hospital (Other)
Other Study IDs: KA 02071
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Infection; Pneumonia; Sepsis; Cross Infection
MeSH Terms: conditions — Infections; Pneumonia; Sepsis; Cross Infection

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Purpose of the study is to investigate and quantify known and possible new riskfactors for nosocomiel infection and death in the intensive care setting.

As new riskfactors Mannose Binding Lechtin and Procalcitonin are chosen and compared to established riskfactors.

ELIGIBILITY:
Inclusion Criteria:Admission to ICU -

Exclusion Criteria:Absence of informed consent and age less than 18 years

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 549
Dates: Start 2002-12; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Dorthe H Olsen, M.D., Principal Investigator — Department of Intensive Care, Herlev University Hospital
Locations (1):
- Department of Intensive Care, Copenhagen, Copenhagen Couty, Denmark